CLINICAL TRIAL: NCT02278861
Title: Low Dose Oral Isotretinoin Versus Topical Tretinoin for Prevention of Actinic Keratosis in Immunocompetent Patients: a Randomized, Comparative Trial
Brief Title: Oral Isotretinoin Versus Topical Tretinoin for Actinic Keratosis
Acronym: ARISOAK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Theraskin (Unknown); Germed Pharma (Industry)
Responsible Party: Principal Investigator, Mayra Ianhez, Assistant Professor, MD, MsC, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UFG 133/11
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Actinic Keratosis
Keywords: actinic keratosis; tretinoin; isotretinoin; cryotherapy; sun protection factor; clinical clearance
MeSH Terms: conditions — Keratosis, Actinic | interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral isotretinoin 10mg/day (Active Comparator): Oral isotretinoin 10mg/day for 6 months The dose could be reduced if there were any significant laboratory alterations or clinical adverse events, along with sunscreen FPS 60 every 3 hours during the day.
  Interventions: Drug: Oral isotretinoin; Drug: Sunscreen FPS 60
- Tretinoin 0,05% cream (Active Comparator): An every other night application of tretinoin 0,05% cream in the face and forearms for 6 months, along with sunscreen FPS 60 every 3 hours during the day.
  If there were any clinical adverse events the drug could be reduced to twice a week.
  Interventions: Drug: Tretinoin 0,05% cream; Drug: Sunscreen FPS 60

INTERVENTIONS:
Drug: Oral isotretinoin — Oral isotretinoin - 10mg/day (one pill) after lunch for six months
  Other Names: Acnova
  Arms: Oral isotretinoin 10mg/day
Drug: Tretinoin 0,05% cream — Topical tretinoin 0,05% cream - applied every other night in the face and forearms for six months
  Other Names: Vitacid 0,05% cream
  Arms: Tretinoin 0,05% cream
Drug: Sunscreen FPS 60 — Sunscreen FPS 60 applied on sun exposed areas every 3 hours daily
  Other Names: Skin Block 60 Fluide Extreme

SUMMARY:
Actinic keratosis (AKs) are premalignant disorders that can evolve into skin cancer. To prevent their development, a study is being conducted with oral isotretinoin and topical tretinoin to verify what drug is the most effective and has the best security profile for these patients. Along with these treatments, cryotherapy with liquid nitrogen and sunscreens will be part of the treatment. The study will have the duration of 10 months. In the first four months, the AKs will be counted and treated with cryotherapy (face and arms) and sunscreens FPS 60 will be used. After it, the patients will return (the AKs will be counted), a new session of cryotherapy will be performed and they will be randomized into two groups: one group using oral isotretinoin 10mg/day ( ISO: 30 patients) and the other one using tretinoin 0,05% cream (AR: 30 patients) applied on face and arms. Skin biopsies will be done for all 60 patients at the beginning of the treatment with retinoids (isotretinoin and tretinoin). After six months of treatment with retinoids, the study will be stopped, AKs will be counted again and skin biopsies will be done. Patients in the group ISO (oral isotretinoin) also have to make blood tests at the beginning, two months and after six months of the treatment. Clinical (AK counting), histological (improvement of parts of the skin) and immunohistochemical parameters will be evaluated to see what drug is more effective for prevention of AKs.

DETAILED DESCRIPTION:
This study is a randomized controlled trial with 60 men and women (already in menopause for at least one year), aged 50-75 years. At the beginning, the number of actinic keratosis (AKs) of face and forearms will be counted and treated with cryotherapy with liquid nitrogen (LN).The patients will be randomized in two groups: one receiving oral isotretinoin 10mg/day every day and other receiving tretinoin 0,05% cream applied in the face and arms every other night, for six months. Along with these treatments, patients will use sunscreens FPS 60 with UVA and UVB protection. The inclusion criteria will be the presence of at least 10 and maximum 40 AKs (visible or palpable). Skin biopsies will be performed twice (before and after treatment with retinoids) for all patients, in the left forearm at a standardized site. Histological and immunohistochemical with blinded- evaluator analysis will be done. The main objective of the study is to evaluate clinical, histological and immunohistochemical effects of retinoids for AK prevention on face and forearms of immunocompetent individuals. Efficacy evaluation will be measured by improving clinical (AK counting before and after treatments), histopathological (Hematoxilin-eosin and Verhoeff staining) and immunohistochemical parameters (markers for carcinogenesis - p53 protein, Bcl-2 and Bax). The secondary objective is evaluate the tolerability and safety of the drugs and their impact in quality of life. The safety analysis will be related to adverse events of the two drugs and the blood tests will be performed in the ISO group patients. Indirectly, by decreasing the number of AKs and the expression of cutaneous carcinogenesis markers, a decrease in the risk of squamous cell carcinoma could be infered . This principle is used by many drugs called chemoprophylactic drugs, and the retinoids are considered in this group.

ELIGIBILITY:
Inclusion Criteria:

1. Signature of the Free and Clarified Consent Term before any procedure of the study;
2. Men and women, aged 50-75 years, in good health;
3. Women in menopause for 1 year or more;
4. Phototypes I-IV by Fitzpatrick classification;
5. Glogau photodamage classification scale from moderate to severe
6. At least 10 and maximum 60 visible and/or palpable actinic keratosis, in the face and forearms, in a standardized distribution;
7. Absence of topical treatment in the face and forearms, except sunscreens, with:

   * tretinoin in the last 6 months;
   * alphahydroxyacids, polyhydroxyacids, betahydroxyacids and ascorbic acid in the last 3 months;
   * drugs or procedures that may change the natural evolution of actinic keratosis, such as imiquimod 5% cream, diclofenac 3% in hyauronic acid gel, photodynamic therapy, 5-FU, in the last 6 months;
8. Absence of previous treatment in the face and forearms with chemical peels and microdermabrasion, in the last 6 months;
9. Absence of previous treatment with oral retinoids in the last 6 months;
10. Absence of anti-cancer chemotherapy in the last 3 months;
11. Absence of hypersensitivity to parabens (present in the majority of drugs as a preserving agent);
12. Absence of infectious or inflammatory diseases in the face and forearms;
13. Absence of immunossupression;
14. Absence of photodermatosis;
15. Agreement in avoiding sun exposure during the research;
16. Agreement in not performing any other kind of treatment that could change the natural history of actinic keratosis; and
17. Agreement with the study conditions, ability to understand and follow strictly the given orientations, availability to attend the periodical evaluations.

For the isotretinoin group (ISO):

1. Absence of history of isotretinoin hypersensitivity;
2. Avoid alcohol intake and;
3. Absence of previous and actual history of rheumatologic diseases.

For the tretinoin group (AR):

1. Absence of history of tretinoin hypersensitivity;

Exclusion Criteria:

For all patients:

1. Men and women who dón't agree with the terms of the research or without ability to understand and/or follow strictly the conditions of the study, without availability to understand and attend the periodical evaluations or who decline to sign the Free and Clarified Consent Term;
2. Patients with less than 10 and more than 60 actinic keratosis in the face and forearms;
3. Fertile, pregnant or lactating women;
4. Fitzpatrick phototypes V e VI ;
5. Topical treatment in the face and forearms, except sunscreens, with:

   * tretinoin in the last 6 months;
   * alphahydroxyacids, polyhydroxyacids, betahydroxyacids and ascorbic acid in the last 3 months;
   * drugs or procedures that may change the natural evolution of actinic keratosis, such as imiquimod 5% cream, diclofenac 3% in hyauronic acid gel, photodynamic therapy, 5-FU, in the last 6 months;
6. Previous treatment in the face and forearms with chemical peels and microdermabrasion, in the last 6 months;

8. Previous treatment with oral retinoids in the last 6 months

For the isotretinoin group (ISO):

1. Presence of significative hepatic laboratory alterations (elevated liver enzymes twice ashigh as the upper normal limit;
2. Diabetic patients, with fast glucose values superior to 110mg/dl;
3. Significant lipid profile alterations (triglycerides > 300 mg/dl; total cholesterol> 250 mg/dl);
4. Low count of white blood cells (leukocytes < 3000/mm3);
5. History of hypersensitivity to isotretinoin and parabens;
6. Alcohol intake;
7. Previous or actual history of rheumatologic diseases;
8. Anticancer chemotherapy in the last 3 months;
9. Previous history of hypervitaminosis A;
10. Previous history of bone or muscular diseases;
11. Patients who are in use or may use the following drugs (risk of drug interaction):

    * tetracyclines and derivatives - in the last 7 days;
    * vitamin A - in the last 30 days;
    * carbamazepine - in the last 7 days.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Reduction in the counting of actinic keratosis in the face and forearms | at the beginning (T0), 120 days (T120) and 300 days (T300)
  The actinic keratosis (AKs) will be counted by the same evaluator twice, in different moments at the same day, at the beginning of the study, after 4 months and at the end (10 months)

SECONDARY OUTCOMES:
Reduction in the thickness of the stratum corneum | 4 months (T120) and 10 months (T300) of the study
  Skin biopsies will be taken from patients at the time of randomization (T120) and after the treatment with retinoids (T300) and stained with hematoxilin-eosin (HE)
Increase in the epithelium thickness | 4 months (T120) and 10 months (T300) of the study
  Skin biopsies will be taken from patients at the time of randomization (T120) and after the treatment with retinoids (T300) and stained with hematoxilin-eosin (HE)
Reduction in the expression of p53 protein | 4 months (T120) and 10 months (T300) of the study
  Skin biopsies will be taken from patients at the time of randomization (T120) and after the treatment with retinoids (T300). Retinoids are known to reduce the expression of this marker of carcinogenesis.
Reduction in the expression of the Bcl-2 protein | 4 months (T120) and 10 months (T300) of the study
  Skin biopsies will be taken from patients at the time of randomization (T120) and after the treatment with retinoids (T300). Retinoids are known to reduce the expression of this marker of carcinogenesis.
Increase in the expression of Bax protein | 4 months (T120) and 10 months (T300) of the study
  Skin biopsies will be taken from patients at the time of randomization (T120) and after the treatment with retinoids (T300). Retinoids are known to increase the expression of this marker of carcinogenesis.

OTHER OUTCOMES:
Reduction in the Dermatology Life Quality Index (DLQI) | at the beginning, with 4 months (T120) and 10 months (T300) of the study
  The Dermatology Life Quality Index (DLQI) questionnaire is performed for every patient at the time frames specified. With the reduction of actinic keratosis and use of retinoids it is expected for retinoids to reduce points of the questionnaire.
Clinical adverse events of tretinoin | 4 months (T120) and 10 months (T300) of the study
  The clinical adverse events with tretinoin 0,05% cream are: erythema, burning sensation, desquamation, irritation The clinical adverse events with oral isotretinoin are: cheilitis, xerophthalmia, xerostomia, dry skin, epistaxis, and other mucocutaneous side effects
Laboratory alterations in patients treated with low dose oral isotretinoin (10mg/day) | 4 months (T120), 6 months (T180) and 10 months (T300). If there were alterations, the laboratory tests were done monthly
  At day 120 (4 months) the patients of isotretinoin group (ISO) were submitted to laboratory tests: complete blood count, alanine and aspartate aminotransferase, fasting plasma glucose test and lipid profile tests.
  At day 180 (6 months) the laboratory tests were repeated, except fasting plasma glucose test At day 300 (10 months) the laboratory tests were asked and repeated after 1 month, except fasting plasma glucose test

CONTACTS AND LOCATIONS:
Overall Officials: Edileia Bagatin, MD, PhD, Study Chair — Federal University of São Paulo UNIFESP; Hélio A Miot, MD, PhD, Study Chair — University of Paulista State - Julio de Mesquita Filho, UNESP
Locations (1):
- Dermatology Outpatient Clinic - Hospital das Clínicas - Federal University of Goias (UFG), Goiânia, Goiás, Brazil

REFERENCES:
- [Result] Ianhez M, Fleury LF Jr, Miot HA, Bagatin E. Retinoids for prevention and treatment of actinic keratosis. An Bras Dermatol. 2013 Jul-Aug;88(4):585-93. doi: 10.1590/abd1806-4841.20131803. PMID 24068130
- [Result] Weinstock MA, Bingham SF, Cole GW, Eilers D, Naylor MF, Kalivas J, Taylor JR, Gladstone HB, Piacquadio DJ, DiGiovanna JJ. Reliability of counting actinic keratoses before and after brief consensus discussion: the VA topical tretinoin chemoprevention (VATTC) trial. Arch Dermatol. 2001 Aug;137(8):1055-8. PMID 11493098